CLINICAL TRIAL: NCT06408116
Title: Predicting Esophageal Cancer Borders Using PET-Imaging PEGASUS
Brief Title: Predicting Esophageal Cancer Borders Using PET-Imaging
Acronym: PEGASUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department head, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-PEGASUS-2023
Record Dates: First submitted 2024-01-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Esophagus Cancer, Stage I; Esophagus Cancer, Stage II
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Photons; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1, Surgery (Other): cT1-2 N0, all histologies: primary surgical therapy
  Interventions: Procedure: surgical therapy
- Group 2, Chemotherapy and surgery (Other): cT3-4 and/or N+, adenocarcinomas: neoadjuvant chemotherapy, surgical therapy
  Interventions: Procedure: surgical therapy; Drug: Chemotherapy
- Group 3, chemotherapy, radiotherapy and surgery (Other): cT3-4 and/or N+, squamous cell carcinomas: neoadjuvant radio(chemo)therapy, surgical therapy
  Interventions: Radiation: photon; Procedure: surgical therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: photon — radiation with 4-5 cm safte margin
  Arms: Group 3, chemotherapy, radiotherapy and surgery
Procedure: surgical therapy — surgery based on PET-CT/MRI staging
Drug: Chemotherapy — neoadjuvant chemotherapy
  Arms: Group 2, Chemotherapy and surgery; Group 3, chemotherapy, radiotherapy and surgery

SUMMARY:
The study examines the diagnostic precision of endosonography, mpMRI and PET/CT in defining tumor boundaries and tumor spread before and after neoadjuvant therapy and definitive surgery.

DETAILED DESCRIPTION:
In Germany, around 7,100 people develop esophageal cancer every year. The treatment of esophageal cancer depends on the histology in addition to the location and tumor stage. Squamous cell carcinomas are differentiated from adenocarcinomas. Until distant metastases are present in functionally operable patients, the treatment of esophageal cancer includes a curative approach using surgical resection with, depending on the risk profile, neoadjuvant chemotherapy or neoadjuvant radio(chemo)therapy. In patients who are functionally inoperable or who refuse surgery, definitive radio(chemo)therapy is given. While the histopathological frozen section is available for surgical resection to differentiate tumor tissue from healthy tissue in addition to the surgeon's macroscopic impression, this assistance in defining the target volume is missing in radiation oncology. Instead, the target volume definition is based, in addition to the contrast-enhanced CT image, on a pretherapeutic endoscopic marking of the tumor boundaries. This allows the tumor boundaries to be delineated in radiation planning imaging. In order to detect the potential microscopic and lymphonodal tumor spread, a large target volume is necessary as a safety margin to avoid later field edge recurrences. According to the current standard, this safety distance extends 4-5cm in both cranial and caudal directions beyond the actual tumor findings. Due to the close positional relationships in the mediastinum, this procedure leads to radiation exposure and subsequent toxicity to the surrounding risk organs such as the lungs, heart and spinal cord. The aim of the present study is to correlate the preoperative endosonographic and imaging local tumor extension and lymph node involvement with the histopathological tumor extension and, in the case of neoadjuvant treatment, with the treatment response by using modern imaging of the tumor and the tumor microenvironment in patients with operated esophageal carcinoma. Since there cannot be any information about the histological tumor extent as a gold standard in the case of definitive radiotherapy, the data from operated patients obtained in the study are extrapolated to the patient population of definitive radiotherapy. From these data, hypotheses should be generated about which patient (groups) benefit from a reduction in the target volume in the definitive radiotherapy treatment setting and whether modern multimodal imaging is suitable for monitoring the therapy response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus, including AEG I and AEG II tumors in the primary situation
* Planned surgical treatment of esophageal carcinoma
* Possible staging advantage through FAPI PET/CT diagnostics
* Patient information and written consent

  -> KI 60% or ECOG 0/1 (at least: self-sufficiency)
* Age ≥ 18 years

Exclusion Criteria:

* Previous radiation therapy in the tumor region
* Previous tumor disease with < 5 years of remission
* Surgical therapy is not functionally or technically possible
* Distant metastasis
* Patient is not capable of giving consent
* Concurrent participation in another clinical trial that could affect the results of this trial or the other trial
* Illnesses that do not allow the person concerned to assess the nature and scope as well as possible consequences of the clinical study
* pregnant or breastfeeding women
* Signs that the person taking part is unlikely to comply with the therapy (e.g. unwillingness to cooperate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Tumor expansion | Before the start of therapy an immediately after the therapy
  Number of patients with correlation of tumor expansion measured by histopathology and imaging techniques (Pet-CT)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No